CLINICAL TRIAL: NCT01337219
Title: Pharmacokinetic Bioequivalence Study of Nebcinal® 150mg/3ml Administered by Aeroneb® Idehaler® Versus Tobi® 300mg/5ml Administered by Pari LC Plus® /Pulmoaide® in Patients With Cystic Fibrosis.
Brief Title: Pharmacokinetic Bioequivalence Study of Nebcinal® 150mg/3ml Administered by Aeroneb® Idehaler® Versus Tobi® 300mg/5ml Administered by Pari LC Plus® /Pulmoaid® in Patients With Cystic Fibrosis
Acronym: RM/NEB-03-10
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Erempharma (Industry)
Collaborators: University of Lyon (Other); Epidemiologie Pharmacologie Investigation Clinique Information medicale Mere Enfant (EPICIME) (Unknown); Clininfo S.A. (Industry); Hospices Civils de Lyon (Other)
Responsible Party: Erempharma, Erempharma
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: RM/NEB-03-10
Record Dates: First submitted 2011-04-13; First posted 2011-04-18 (Estimated); Last update posted 2011-04-18 (Estimated); Status verified 2011-02

CONDITIONS: Cystic Fibrosis
Keywords: cystic fibrosis; bioequivalence; pharmacokinetic; sputum; plasma
MeSH Terms: conditions — Cystic Fibrosis | interventions — Tobramycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm A (Other): experimental treatment (Nebcinal/Aeroneb Idehaler pocket) - 6day-wash out period - standard treatment (Tobi/Pari LC Plus)
  Interventions: Drug: Tobramycin
- Arm B (Other): standard treatment (Tobi/Pari LC Plus) - 6day-wash out period - experimental treatment (Nebcinal/Aeroneb Idehaler)
  Interventions: Drug: Tobramycin

INTERVENTIONS:
Drug: Tobramycin

SUMMARY:
Cystic fibrosis (CF) is a genetic disease characterized by mutations in CFTR (Cystic Fibrosis Transmembrane conductance Regulator) gene. Mortality and morbidity are mostly related to the respiratory affection which appears early in neonates.

The constant improvement in symptomatic treatments and care strategies allowed CF patients' life expectancy to be increased over the last decades.

Vital prognostic is related to bronchopulmonary infections. 39% of CF patients under 18 years old and 70% of adult CF patients are chronically infected by Pseudomonas aeruginosa.

Elevated concentrations of tobramycin in broncho secretions, about 1000 times the MIC, is obtained by inhaled administration of tobramycin and is active against in-vitro resistant Pseudomonas aeruginosa.

Study hypotheses :

Regarding literature data and in-vitro studies, the administration of Nebcinal® 150mg/3ml administered twice a day by Aeroneb® Idehaler® pocket® would deliver the same quantity of antibiotic in lung and plasma as Tobi® 300mg/5ml administered twice a day by Pari® LC Plus® in children and adult patients with CF.

Primary objective :

To compare plasma concentrations after inhalation of Nebcinal® 150mg/3ml administered by Aeroneb® Idehaler pocket® and Tobi® 300 mg/5ml administered by Pari LC Plus®

ELIGIBILITY:
Inclusion Criteria:

* Adults and children aged 6 years old and more
* Male or female
* Patients with cystic fibrosis (positive sudoral test, Cl > 60 mmol/L)
* Followed in a CRCM (CF care centre)
* FEV1 ≥40%
* Informed consent collected from adults or parents or legal guardians and children.
* Affiliation to the National Health Insurance program (Sécurité sociale).

Exclusion Criteria:

* renal insufficiency defined by a creatinine clearance level superior to 2 mg/dl
* recent pneumothorax, emphysema, punction or recent pleural biopsy, recent haemoptysis superior to 60 ml within 30 days prior to randomization
* Acute pulmonary exacerbation pathology, according to conference of consensus (2002), evaluated by :
* Cough increase
* Sputum increase
* Decrease in tolerance to effort
* Loss of weight, lack of appetite
* Deterioration of respiratory function
* Medical history of intolerance, toxicity or allergy to tobramycin, hypersensitivity to aminoside

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2011-04; Primary Completion 2011-09 (Estimated)

PRIMARY OUTCOMES:
Plasma concentration of tobramycin from 0 to 8h after administration | from 0 to 8h after administration

SECONDARY OUTCOMES:
sputum of tobramycin concentrations | from 0 to 8 hours after administration
Safety of Nebcinal® 150mg/3ml administered by Aeroneb® Idehaler pocket®; | 15 days
Time of nebulization of Nebcinal® 150mg/3ml administered by Aeroneb® Idehaler pocket® | during nebulization
Satisfaction of Nebcinal® 150mg/3ml administered by Aeroneb® Idehaler pocket® | after administration of the drug, in average 20 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Gabriel Bellon, Principal Investigator — Centre de Resources et de competences pour la mucovisidose; Isabelle Durieu, Pr, Principal Investigator — Centre de Resources et de competences pour la mucovisidose Hôpital Lyon Sud; behrouz Kassai, Dr, Study Chair — University of Lyon
Locations (1):
- Centre de Ressource et de Compétence Mucoviscidose Pédiatrique Centre de Référence Mucoviscidose, Lyon, France